CLINICAL TRIAL: NCT05444205
Title: The Pittsburgh Study Early Childhood Collaborative
Brief Title: The Pittsburgh Study Early Childhood
Acronym: TPS-ECC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Grable Foundation (Unknown); The Shear Family Foundation (Unknown); Heinz Endowments (Other)
Responsible Party: Principal Investigator, Daniel Shaw, Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY19060235
Record Dates: First submitted 2022-02-25; First posted 2022-07-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Child Development; Child Language; Child Behavior Problem; Parenting; Parent Child Abuse

STUDY DESIGN:
Intervention Model Description: The Early Childhood Collaborative is an implementation study and therefore, all participants are offered intervention. An innovative aspect of the study is supporting parent choice of intervention. Participants are given a choice of interventions based on a tiered model, and they can also decline to engage in programs and continue in follow-up.
Masking Description: The Early Childhood Collaborative is an implementation study and therefore, all participants are offered intervention and there in so masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Higher resources/lower challenges (Experimental): Participants are assigned to this arm based on results of a brief screen; self-reports indicated that they did not posses any measured risk factors. Participants are provided with a choice of the following preventive interventions: Text4Baby/Bright by Text (depending on child age), Nurture Program, and/or Family Centers.
  Interventions: Behavioral: Text4Baby or Bright by Text Referral; Behavioral: Nurture Program Warm Referral; Behavioral: Family Center Warm Referral
- Lower Resources/Lower Challenges (Experimental): Participants are assigned to this arm based on results of a brief screen; self-reports indicated that they were low-income, a teen parent, their newborn had health challenges (more than five weeks premature or a neonatal intensive care unit stay of longer than 4 weeks, or they reported mild parenting challenges. They did not endorse any more serious measured risk factors. Participants are provided with a choice of the following preventive interventions: Nurture Program and/or Video Interaction Project.
  Interventions: Behavioral: Nurture Program Warm Referral; Behavioral: Video Interaction Project
- Moderate Challenges (Experimental): Participants are assigned to this arm based on results of a brief screen; self-reports indicated that they had a history of mental health problems, low social support, or moderate parenting challenges. They did not endorse any more serious measured risk factors. Participants are provided with a choice of the following preventive interventions: Nurture Program and/or Video Interaction Project.
  Interventions: Behavioral: Video Interaction Project; Behavioral: Family Check-UP
- Serious Challenges (Experimental): Participants are assigned to this arm based on results of a brief screen; self-reports indicated that they had a histories of involvement with child welfare, incarceration, opioid use disorder, recent homelessness, or that their child is displaying serious behavior problems. Participants are provided with a choice of the following preventive interventions: Smart Beginnings, Family Check-Up or if the child was less than two weeks old, Healthy Families America.
  Interventions: Behavioral: Family Check-UP; Behavioral: Smart Beginnings; Behavioral: Healthy Families America Warm Referral

INTERVENTIONS:
Behavioral: Text4Baby or Bright by Text Referral — Passive texting programs where participants receive free text messages on topics such as child development and parenting tips three times per week. Text4Baby serves parents of children under one year. Bright by Text serves parents of children under eight years of age.
  Arms: Higher resources/lower challenges
Behavioral: Nurture Program Warm Referral — Nurture Program is a nonprofit organization that promotes healthy development in young children by pairing moms with experienced and knowledgeable mentors who use text messaging to answer questions and provide helpful information, while offering support and encouragement throughout the child's first few years of life.
  Arms: Higher resources/lower challenges; Lower Resources/Lower Challenges
Behavioral: Video Interaction Project — The Video Interaction Project is a program to support parents and their young children. Video Interaction Project is typically offered at a convenient location, such as a pediatric clinic. Parents are observed and videotaped for 3 to 5 minutes while interaction with their child. The Video Interaction Project coach then watches the video with the parent and talks about their interaction, highlighting how best to support the child's growth and language development.
  Arms: Lower Resources/Lower Challenges; Moderate Challenges
Behavioral: Family Check-UP — The Family Check-Up is brief, taking place over the course of three sessions, each about an hour long. A Family Check-Up family coach will spend time getting to know the family during an "Initial Interview." Second, parents complete questionnaires that assess child and family adjustment, relationships, and other areas that influence children and families. The assessment includes videotaped family interaction tasks, where parents take part in activities with their child like playing together with toys and puzzles. Third, the Feedback session consists of sharing feedback - including strengths and challenges - about child and family well-being based on survey responses and video clips. Parents are invited to set goals for their family to support and maintain strengths and address areas of concern. Parents are paid 25 dollars after the Feedback Session. Parents have the option to continue meeting with the family coach to support the child's development and improve parental well-being.
  Arms: Moderate Challenges; Serious Challenges
Behavioral: Smart Beginnings — Smart Beginnings consists of delivering both Video Interaction Project and the Family Check-up packed together as a single intensive intervention.
  Arms: Serious Challenges
Behavioral: Healthy Families America Warm Referral — As part of Healthy Families America, professionally trained Nurse Home Visitors provide information during weekly home visits so that parents can provide the best for your new baby. Topics addressed are ways to keep the baby safe, how to take care of the baby, and activities parents can enjoy with their babies.
  Arms: Serious Challenges
Behavioral: Family Center Warm Referral — There are 27 Family Centers across Allegheny County provide services to families of young children 5 and under. These centers focus on three primary activities: 1. enhancing child development; 2. facilitating parent education, and 3. ensuring parents are supported and connected.
  Arms: Higher resources/lower challenges

SUMMARY:
The Early Childhood Collaborative of The Pittsburgh Study is a community-partnered, county-wide implementation of programs for children and families from birth through formal school entry to address real-world challenges that exist in providing effective preventive interventions for families with young children, particularly low-income families.

DETAILED DESCRIPTION:
The Early Childhood Collaborative of The Pittsburgh Study is a community-partnered, county-wide implementation of programs for children and families from birth through formal school entry to address real-world challenges that exist in providing effective preventive interventions for families with young children, particularly low-income families. Specifically, The Early Childhood Collaborative seeks to increase engagement (uptake and retention) in evidence-based interventions by (1) initially assessing families' resources and challenges, (2) offering families a menu of intervention options tailored to their resources/needs, and (3) providing these services at multiple locations to optimize accessibility. The Early Childhood Collaborative involves population-level utilization of multiple platforms that families, particularly families at greater risk for health disparities, typically use, including health care (birthing hospitals, pediatric care, federally qualified health centers), Women, Infants, and Children nutritional clinics, and family centers. The Early Childhood Collaborative will locate services in these platforms and at family's homes. The Early Childhood Collaborative focuses on child thriving and flourishing as key outcomes of interest, and community strengths as key drivers of change. To promote sustainability, investigators include representatives from the Departments of Human Services and Health who are responsible for funding and implementing home visiting programs in the greater Pittsburgh community, with the goal of generating infrastructures and capacity in existing community agencies for providing evidence-based behavioral health care.

ELIGIBILITY:
Inclusion Criteria:

* Allegheny County Residency, legal custodian of child

Exclusion Criteria:

* Non-English speaking

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24000 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Child inhibitory control | 4 years
  Change in inhibitory control as measured using the 13-item Inhibitory Control scale of the Children's Behavior Questionnaire. Mean scores will be calculated with a possible range of 0-7 (higher scores indicate greater inhibitory control).
  Citation: Rothbart, M. K., Ahadi, S. A., Hershey, K. L. & Fisher, P. (2001). Investigations of temperament at 3-7 years: The Children's Behavior Questionnaire. Child Development, 72(5), 1394-1408.
Parent Reading Behaviors - Infancy | 4 years
  Change in parent reading behaviors as measured using the StimQ self-report. We will use the 15-item reading factor. Scores used for outcome will be determined by our collaborator (and scale developer) Dr. Alan Mendelsohn and his research team at NYU.
  Citations:
  StimQ2-Infant©2016. NYU School of Medicine Alan L. Mendelsohn MD, Carolyn B. Cates PhD, Matthew Johnson, PhD, Adriana Weisleder PhD, Benard Dreyer MD
Socioemotional adjustment - ITSEA | 4 years
  Change in infant and toddler problem behaviors and socioemotional adjustment: Measured by the The infant-toddler social and emotional assessment (ITSEA). We will use the 14-item negative emotionality factor. Items are measured on a 3-point likert-type scale. A sum score will be calculated, with a possible range of 0-28 (higher scores indicate greater problems).
  Citations: Carter, A. S., Briggs-Gowan, M. J., Jones, S. M., & Little, T. D. (2003). The infant-toddler social and emotional assessment (ITSEA): Factor structure, reliability, and validity. Journal of abnormal child psychology, 31(5), 495-514.
Socioemotional adjustment - BITSEA | 4 years
  Change in infant and toddler problem behaviors: Measured by a subset of 28 items derived from the Brief infant-toddler social and emotional assessment (BITSEA) Total Problems scale. Items are measured on a 3-point likert-type scale. A sum score will be calculated, with a possible range of 0-56 (higher scores indicate greater problems).
  Citation: Briggs-Gowan, M. J. & Carter, A.S. (2006). BITSEA : Brief infant-toddler social and emotional assessment. San Antonio, TX: Pearson 2006.
Socioemotional adjustment - CBCL | 4 years
  Change in child problem behaviors and socioemotional adjustment: Measured by the Child Behavior Checklist (CBCL). We will use 60 items that comprise the Externalizing and Internalizing broadband factors. Items are measured on a 3-point Likert-type scale. A raw sum score will be calculated for each factor, with a possible range of 0-48 for Externalizing problems and 0-72 for Internalizing problems (higher scores indicate greater problems). We will also calculate t-scores for both scales.
  Citation: Achenbach, T. M. (2009). The Achenbach System of Empirically Based Assessment (ASEBA): Development, Findings, Theory, and Applications. Burlington, VT: University of Vermont Research Center for Children, Youth, & Families.

SECONDARY OUTCOMES:
Positive parenting skills - PYB | 4 years
  Change in proactive and positive parenting strategies for parents of infants as measured by Parenting Your Baby (adapted from the Parenting Young Children measure cited below). The measure is comprised of an 8-item positive/supportive parenting score and a 5 item proactive parenting score. Mean scores will be calculated with a possible range of 1-7. Higher scores indicated positive parenting skills.
  Citation: McEachern, A.D., Dishion T.D., Weaver, C.M., Shaw, D.S., Wilson, M N. & Gardner, F. (2011). Parenting Young Children (PARYC): Validation of a self-report parenting measure. Journal of Child and Family Studies, 1-14.
Positive parenting skills - PYT | 4 years
  Change in proactive and positive parenting strategies for parents of toddlers as measured by Parenting Your Toddler (adapted from the Parenting Young Children measure cited below). The measure is comprised of a 7-item positive/supportive parenting score, a 7-item proactive parenting score, and 7-items limit setting score. Mean scores will be calculated with a possible range of 1-7. Higher scores indicate positive parenting skills.
  Parenting Young Children. Citation: McEachern, A.D., Dishion T.D., Weaver, C.M., Shaw, D.S., Wilson, M N. & Gardner, F. (2011). Parenting Young Children (PARYC): Validation of a self-report parenting measure. Journal of Child and Family Studies, 1-14.
Positive parenting skills - PARYC | 4 years
  Change in proactive and positive parenting strategies as measured by Parenting Young Children. The measure is comprised of a 7-item positive/supportive parenting score, a 7-item proactive parenting score, and 7-items limit setting score. Mean scores will be calculated with a possible range of 1-7. Higher scores indicate positive parenting skills.
  Citation: McEachern, A.D., Dishion T.D., Weaver, C.M., Shaw, D.S., Wilson, M N. & Gardner, F. (2011). Parenting Young Children (PARYC): Validation of a self-report parenting measure. Journal of Child and Family Studies, 1-14.
Harsh parenting | 4 years
  Change in harsh parenting strategies as measured by the 5-item Harsh Parenting Scale. Items are measured on a 6-point Likert-type scale. A sum score will be calculated, with a possible range of 5-30. Higher scores indicate harsher parenting.
  Citation: Socolar, R. R. S. & Stein, R. E. K. (1995). Spanking Infants and Toddlers: Maternal Belief and Practice. Pediatrics, 95, 105-111.
Parent depressive symptoms | 4 years
  Change in depressive symptoms as measured by the 20-item Centers for Epidemiological Studies-Depression (CES-D). Items are measured on a 4-point Likert-type scale. A sum score will be calculated, with a possible range of 0-60. Higher scores indicate higher levels of depressive symptoms. Note this measure has a clinical cut-off of 16 meaning that scores greater than or equal to 16 indicate clinically significant levels of depression.
  Citation: Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Applied Psychological Measurement. 1977;1:385-401.
Parent anxiety symptoms | 4 years
  Change in parent anxiety symptoms as measured by the GAD-7. Items are measured on a 4-point Likert-type scale. A sum score will be calculated, with a possible range of 0-21. Higher scores indicate higher levels of anxiety symptoms.
  Citation: Spitzer, R.L., Kroenke, K., Williams, J.B.W., Lowe, B. (2006). A brief measure for assessing generalized anxiety disorder. Archives of Internal Medicine,166,1092-1097.
Parent social support | 4 years
  Change in social support as measured by the 3-item social support subscale of the Comprehensive Inventory of Thriving. Items are measured on a 5-point Likert-type scale. A sum score will be calculated, with a possible range of 3-15. Higher scores indicate greater social support.
  Citation: Su, R., Tay, L., & Diener, E. (2014). The development and validation of Comprehensive Inventory of Thriving (CIT) and Brief Inventory of Thriving (BIT). Applied Psychology: Health and Well-Being. Published online before print. doi: 10.1111/aphw.12027
Well-child care | 4 years
  Change in well-child pediatric visits and receipt of immunizations. Measured by medical records released by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, PhD, Study Director — University of Pittsburgh
Locations (5):
- United States (5):
  - Primary Care Health Services, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh Primary Care Centers, Pittsburgh, Pennsylvania
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Allegheny County Family Centers, Pittsburgh, Pennsylvania
  - Women, Infants, and Children Program, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be made public after the trial.
Supporting Information: Study Protocol
Time Frame: De-identified data will be made public at the conclusion of the study. The data will be available indefinitely.
Access Criteria: Data will be available to anyone who wishes to access the data for any type of analysis.

REFERENCES:
- [Derived] Krug CW, Mendelsohn AL, Wuerth J, Roby E, Shaw DS. The Pittsburgh Study: A Tiered Model to Support Parents during Early Childhood. J Pediatr. 2025 Feb;277:114396. doi: 10.1016/j.jpeds.2024.114396. Epub 2024 Nov 12. PMID 39536860
- See also: The Pittsburgh Study website — https://thepittsburghstudy.org/